CLINICAL TRIAL: NCT06228677
Title: Comparison of Catecholamine Concentrations in Adrenal Venous Blood and Peripheral Venous Blood During Percutaneous Selective Adrenal Artery Embolization in Hypertensive Patients With Primary Aldosteronism: A Prospective Cohort Study
Brief Title: Comparison of Catecholamine Concentrations in Venous Blood During Selective Adrenal Artery Embolization
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: CCC-SAAE
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Resistant Hypertension; Secondary Hypertension; Secondary Hypertension to Endocrine Disorders; Primary Aldosteronism
Keywords: Primary Aldosteronism; Selective Adrenal Artery Embolization; catecholamine concentration; Adrenal Venous Blood; Blood Pressure Variability
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adrenal Venous Sampling Group: Adrenal veinous sampling in patients with primary aldosteronism who underwent percutaneous selective adrenal artery embolization
  Interventions: Procedure: Selective adrenal artery embolization
- Peripheral Venous Sampling Group: Peripheral veinous sampling in patients with primary aldosteronism who underwent percutaneous selective adrenal artery embolization
  Interventions: Procedure: Selective adrenal artery embolization

INTERVENTIONS:
Procedure: Selective adrenal artery embolization — Percutaneous selective adrenal artery embolization in patients with primary aldosteronism

SUMMARY:
To explore the relationship between perioperative blood pressure and catecholamine concentrations in adrenal venous blood and peripheral venous blood in hypertensive patients with primary aldosteronism (PA) who underwent percutaneous selective adrenal artery embolization (SAAE). In order to elucidate the related phenomena and possible mechanisms of blood pressure fluctuations caused by SAAE treatment in hypertensive patients with PA.

DETAILED DESCRIPTION:
Percutaneous selective adrenal artery embolization (SAAE) is a minimally invasive interventional procedure that allows for necrosis of diseased adrenal glands by selectively embolizing the adrenal arteries supplying the lesion using an embolic agent to block the overproduction of aldosterone, and has been used as a treatment for PA as a minimally invasive alternative. However, it is of concern that in our team's SAAE practice, we have found that some patients with PA experience a dramatic increase in blood pressure during surgery, even exceeding 220/130 mmHg, yet some patients do not experience significant fluctuations in blood pressure. The perioperative risk is undoubtedly significantly increased for patients with high blood pressure fluctuations. What are the reasons for this discrepancy phenomenon? Therefore, the present study was designed to synchronize adrenal vein blood collection in PA hypertensive patients undergoing SAAE, and to compare the perioperative adrenal vein blood and peripheral venous blood catecholamine concentrations, with a view to discovering the patterns and possible causes of blood pressure fluctuations, hormone level changes, and other phenotypic changes, and elucidating the possible mechanisms of blood pressure fluctuations triggered by SAAE treatment of PA hypertension, in order to provide an evidence-based basis for minimally invasive interventional therapy for PA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years with no gender restrictions.
2. Adherence to the "Primary Aldosteronism" Diagnosis and Treatment Guidelines, confirmed diagnosis of primary aldosteronism following rigorous drug washout, and identification as either aldosteronoma or idiopathic aldosteronism via adrenal vein blood sampling.
3. Blood pressure metrics that satisfy any of the subsequent conditions: a) Clinic-recorded blood pressure ≥140/90mmHg; b) 24-hour ambulatory blood pressure monitoring results displaying average blood pressure >130/80 mmHg or daytime readings >135/85 mmHg.
4. Adrenal CT scan revealing adrenal hyperplasia, nodular formations, or no significant morphological deviations.
5. Hypertension history surpassing a duration of 6 months.
6. Prior to screening, patients or their lawful guardians must provide a signed informed consent, sanctioned by the ethics committee.

Exclusion Criteria:

1. Patients diagnosed with primary hypertension or secondary hypertension attributed to other etiologies.
2. Female participants who are presently pregnant, lactating, or with intentions to conceive within the forthcoming year.
3. Presence of significant systemic diseases, with particular attention to hepatic and renal dysfunction.
4. Pronounced allergic reaction to contrast agents.
5. Any other serious systemic diseases with a life expectancy of less than 12 months.
6. Participants concurrently enrolled or expressing interest to participate in other clinical trials, the outcomes of which could potentially influence the results of the current study.
7. The researcher's discretion deems the subject inappropriate for inclusion in the study for any given reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients with a definite diagnosis of primary aldosteronism who agree to undergo percutaneous selective adrenal artery embolization.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Invasive blood pressure | Selective adrenal artery embolization immediately, after 5 minutes, 15 minutes, 30 minutes
  Auxiliary check
24-hour dynamic blood pressure | Selective adrenal artery embolization before 24 hours, after 24 hours
  Auxiliary check
Plasma Norepinephrine | Selective adrenal artery embolization immediately, after 5 minutes, 15 minutes, 30 minutes
  Biochemical indicators
Plasma Adrenaline | Selective adrenal artery embolization immediately, after 5 minutes, 15 minutes, 30 minutes
  Biochemical indicators
Plasma Dopamin | Selective adrenal artery embolization immediately, after 5 minutes, 15 minutes, 30 minutes
  Biochemical indicators
Plasma Renin | Selective adrenal artery embolization immediately, after 5 minutes, 15 minutes, 30 minutes
  Biochemical indicators
Plasma Aldosterone | Selective adrenal artery embolization immediately, after 5 minutes, 15 minutes, 30 minutes
  Biochemical indicators
Serum sodium | Selective adrenal artery embolization immediately, after 5 minutes, 15 minutes, 30 minutes
  Biochemical indicators
Serum potassium | Selective adrenal artery embolization immediately, after 5 minutes, 15 minutes, 30 minutes
  Biochemical indicators

CONTACTS AND LOCATIONS:
Overall Officials: Peijian Wang, PhD, Principal Investigator — First Affiliated Hospital of Chengdu Medical College
Locations (1):
- The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Shared with the researchers' consent
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year after the research is completed and the results are published.
Access Criteria: Via the corresponding author's email

REFERENCES:
- [Background] Stavropoulos K, Imprialos KP, Patoulias D, Katsimardou A, Doumas M. Impact of Primary Aldosteronism in Resistant Hypertension. Curr Hypertens Rep. 2022 Aug;24(8):285-294. doi: 10.1007/s11906-022-01190-9. Epub 2022 Apr 21. PMID 35445928
- [Background] Huang WC, Lin YH, Wu VC, Chen CH, Siddique S, Chia YC, Tay JC, Sogunuru G, Cheng HM, Kario K. Who should be screened for primary aldosteronism? A comprehensive review of current evidence. J Clin Hypertens (Greenwich). 2022 Sep;24(9):1194-1203. doi: 10.1111/jch.14558. PMID 36196469
- [Background] Meng Z, Dai Z, Huang K, Xu C, Zhang YG, Zheng H, Liu TZ. Long-Term Mortality for Patients of Primary Aldosteronism Compared With Essential Hypertension: A Systematic Review and Meta-Analysis. Front Endocrinol (Lausanne). 2020 Mar 10;11:121. doi: 10.3389/fendo.2020.00121. eCollection 2020. PMID 32210920
- [Background] Monticone S, D'Ascenzo F, Moretti C, Williams TA, Veglio F, Gaita F, Mulatero P. Cardiovascular events and target organ damage in primary aldosteronism compared with essential hypertension: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2018 Jan;6(1):41-50. doi: 10.1016/S2213-8587(17)30319-4. Epub 2017 Nov 9. PMID 29129575
- [Background] Funder JW, Carey RM. Primary Aldosteronism: Where Are We Now? Where to From Here? Hypertension. 2022 Apr;79(4):726-735. doi: 10.1161/HYPERTENSIONAHA.121.18761. Epub 2022 Jan 24. PMID 35067069
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Lu YC, Liu KL, Wu VC, Wang SM, Lin YH, Chueh SJ, Wu KD, Su YR, Huang KH; TAIPAI Study Group. Unilateral adrenalectomy in bilateral adrenal hyperplasia with primary aldosteronism. J Formos Med Assoc. 2023 May;122(5):393-399. doi: 10.1016/j.jfma.2022.12.015. Epub 2023 Feb 20. PMID 36813699
- [Background] Tezuka Y, Turcu AF. Real-World Effectiveness of Mineralocorticoid Receptor Antagonists in Primary Aldosteronism. Front Endocrinol (Lausanne). 2021 Mar 26;12:625457. doi: 10.3389/fendo.2021.625457. eCollection 2021. PMID 33841329
- [Background] Fowler AM, Burda JF, Kim SK. Adrenal artery embolization: anatomy, indications, and technical considerations. AJR Am J Roentgenol. 2013 Jul;201(1):190-201. doi: 10.2214/AJR.12.9507. PMID 23789675
- [Background] Hokotate H, Inoue H, Baba Y, Tsuchimochi S, Nakajo M. Aldosteronomas: experience with superselective adrenal arterial embolization in 33 cases. Radiology. 2003 May;227(2):401-6. doi: 10.1148/radiol.2272011798. Epub 2003 Apr 3. PMID 12676966
- [Background] Zhao Z, Liu X, Zhang H, Li Q, He H, Yan Z, Sun F, Li Y, Zhou X, Bu X, Wu H, Shen R, Zheng H, Yang G, Zhu Z; Chongqing Endocrine Hypertension Collaborative Team. Catheter-Based Adrenal Ablation Remits Primary Aldosteronism: A Randomized Medication-Controlled Trial. Circulation. 2021 Aug 17;144(7):580-582. doi: 10.1161/CIRCULATIONAHA.121.054318. Epub 2021 Aug 16. No abstract available. PMID 34398686
- [Background] Zhou Y, Liu Q, Wang X, Wan J, Liu S, Luo T, He P, Hou J, Pu J, Wang D, Liang D, Yang Y, Wang P. Adrenal Ablation Versus Mineralocorticoid Receptor Antagonism for the Treatment of Primary Aldosteronism: A Single-Center Prospective Cohort Study. Am J Hypertens. 2022 Dec 8;35(12):1014-1023. doi: 10.1093/ajh/hpac105. PMID 36205513